CLINICAL TRIAL: NCT04164238
Title: Phase II Trial of Neoadjuvant Anti-PD-1 Antibody (Toripalimab) or Combined With Chemotherapy in Head and Neck Squamous Cell Carcinoma Patients
Brief Title: Neoadjuvant Anti-PD-1 Antibody (Toripalimab) or Combined With Chemotherapy in HNSCC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yulong Zheng, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJU20191451
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; PD-1 antibody; Neoadjuvant; Major pathologic response
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab; Paclitaxel; Carboplatin; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Toripalimab 240mg IV, every 3 weeks;
  Interventions: Drug: Toripalimab
- Arm B (Experimental): Toripalimab 240mg IV, Q3W; Paclitaxel 175mg/m^2, IV, Q3W; Carboplatin AUC 5, IV, Q3W
  Interventions: Drug: Toripalimab; Drug: Paclitaxel; Drug: Carboplatin
- Arm C (Experimental): Toripalimab 240mg IV, Q3W; Paclitaxel 175mg/m^2, IV, Q3W; Cisplatin 25mg/m^2 IV,d1-d3, Q3W; 5-FU 3000mg/m^2 CIV 72h, Q3W
  Interventions: Drug: Toripalimab; Drug: Paclitaxel; Drug: Cisplatin; Drug: 5-fu

INTERVENTIONS:
Drug: Toripalimab — Toripalimab Injection
Drug: Paclitaxel — Paclitaxel Injection
  Arms: Arm B; Arm C
Drug: Carboplatin — Carboplatin Injection
  Arms: Arm B
Drug: Cisplatin — Cisplatin injection
  Arms: Arm C
Drug: 5-fu — 5-fu injection
  Arms: Arm C

SUMMARY:
This study evaluate either Toripalimab or combined with chemotherapy as neoadjuvant treatment for patients with head and neck squamous cell carcinoma. Participants in arm A receive Toripalimab, in arm B receive Toripalimab plus PC (paclitaxel and carboplatin), arm C with Toripalimab plus modified TPF(paclitaxel and cisplatin and 5-fu).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pathologic or cytologic diagnosis of squamous cell carcinoma of head and neck;
* Resectable or potentially resectable lesion;
* ECOG PS 0-1;
* Age >18 years old;
* At least one target lesion according to RECIST 1.1;
* Proper function of the cardiovascular system, liver, kidney and bone marrow for receiving chemotherapy and surgery;

Exclusion Criteria:

* Distant metastasis;
* Second malignancy within 5 years;
* Nasopharyngeal carcinoma;
* Active autoimmune diseases;
* HIV infected;
* Required prednisone dose >=10mg daily;
* Heart attack within 6 months;
* Stroke within 6 months;
* Other conditions that investigators consider the patients are not suitable for PD-1antibody;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-11-07 (Estimated); Study Completion 2021-11-07 (Estimated)

PRIMARY OUTCOMES:
MPR | 6 weeks
  major pathologic response

SECONDARY OUTCOMES:
AE | 2 years
  adverse events
RFS | 2 years
  recurrence free survival
ORR | 6 weeks
  overall response rate
PFS | 6 months
  progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Nong Xu, MD, Study Chair — Zhejiang University
Locations (1):
- Department of Medical Onocology, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China